CLINICAL TRIAL: NCT03118817
Title: A Single-arm, Open-label, Multi-center, Phase I Expansion Study Evaluating the Efficacy and Safety of HM95573 Monotherapy in Patients With BRAF, KRAS or NRAS Mutation-positive Solid Cancers
Brief Title: Expansion Study to Evaluate the Efficacy and Safety of HM95573 in BRAF, KRAS or NRAS Mutant Solid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-RAFI-102
Record Dates: First submitted 2017-03-20; First posted 2017-04-18 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HM95573 (Experimental): Single arm
  Interventions: Drug: HM95573

INTERVENTIONS:
Drug: HM95573 — Dose: 450 mg BID
  Regimen: twice daily (BID), continuous dosing
  Duration: until progression disease or unacceptable toxicity develops

SUMMARY:
This study evaluates the anti-tumor efficacy and safety of single agent HM95573 administered in patients with solid tumors harboring mutations in either BRAF, KRAS or NRAS gene.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor
* Confirmed mutations in either BRAF, KRAS or NRAS gene
* Eligible for biomarker analysis as follows:

  * Be able to provide an archival tumor tissue at screening.
  * Consent to undergo pre- and post-treatment tumor biopsies, provided sites of disease are easily and safely accessible
* Tumors for which standard therapy either does not exist or has proven ineffective or intolerable at study entry;
* At least one lesion (excluding brain) measureable per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
* Life expectancy of ≥ 12 weeks;
* ECOG performance status score 0 or 1;
* Adequate organ function

Exclusion Criteria:

* Hematologic malignancy or double primary cancer.
* Treatment with any of the following:

  * Anticancer therapy including chemotherapy, hormonal treatment, or radiotherapy within 14 days of the first dose of study drug.
  * Investigational (not-approved) agent within 28 days or 5 fold of its half-life prior to the first dose of study drug.
  * Major surgical procedure within 28 days prior to the first dose of study drug.
  * Systemic corticosteroid (≥ 10mg prednisolone or equivalent dose of other anti-inflammatory corticosteroids) or systemic immunosuppressant within 28 days prior to the first dose of study drug or current systemic immunosuppressant which is required to be used continuously during treatment period of the study. But following treatments will be allowed: topical applications, inhaled sprays, eye drops, or local injections.
  * Treatment with nitrosourea, mitomycin, ipilimumab or other immunotherapy within 42 days prior to the first administration of study drug.
  * >5 prior anticancer therapy regimens
* Spinal cord compression, leptomeningopathy or other symptomatic or uncontrolled central nervous system or brain metastasis.
* Cardiovascular abnormalities as follow:

  * mean QTcF > 440 msec
  * Heart failure of NYHA Class III or IV
  * Heart metastasis
  * Uncontrolled serum electrolyte disturbances (hyponatremia, hypokalemia, hypocalcemia or hypomagnesemia)
  * History of acute coronary syndrome including unstable angina and myocardial infarction, uncontrolled arrhythmias (except for sinus arrhythmia and atrial fibrillation which is controlled within 30 days prior to the first dose of study drug), symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose of study drug.
  * History of coronary angioplasty, coronary/peripheral artery bypass graft or stent insertion within 6 months prior to the first dose of study drug.
  * History of congenital long QT syndrome or clinically significant ≥ Grade 2 (NCI-CTCAE version 4.03) ventricular or atrial dysrhythmias.
* Ophthalmologic disorders as follows:

  * History of or evidence of retinal vein occlusion (RVO), central serous retinopathy (CSR) or neovascular macular degeneration at screening
  * Glaucoma with intraocular pressure ≥ 21 mmHg

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate (Proportion of patients with reduction in tumor burden of a predefined amount) | At screening and every 8 weeks from time of first dosing until date of progression, start of other anticancer therapy or death whichever came first, assessed up to study completion (around 36 months).

SECONDARY OUTCOMES:
Safety and tolerability by assessing adverse events (AEs) based on CTCAE ver.4.03 | All AEs occurring up to 28 days after the last administration of study drug until the start of other anti-cancer treatment, whichever comes first, will be record.
Best overall response rate | At screening and every 8 weeks from time of first dosing until date of progression, start of other anticancer therapy or death whichever came first, assessed up to study completion (around 36 months).
Disease control rate | At screening and every 8 weeks from time of first dosing until date of progression, start of other anticancer therapy or death whichever came first, assessed up to study completion (around 36 months).
Progression-free survival | At screening and every 8 weeks from time of first dosing until date of progression, start of other anticancer therapy or death whichever came first, assessed up to study completion (around 36 months).
Changes in molecular biomarkers | Screening and 15 days after first dosing

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Korea, Republic of, Gyeonggi-do, Seongnam-si, Gyeonggi-do
  - Korea, Republic of, Gyeongsangbuk-do, Daegu, Gyeongsangbuk-do
  - Korea, Republic of, Chungcheongbuk-do, Cheongju-si, North Chungcheong
  - Korea, Republic of, Seoul, Seoul